CLINICAL TRIAL: NCT04756037
Title: A Phase 3, Single-Arm, Open-Label Study to Evaluate the Safety and Contraceptive Efficacy of Relugolix Combination Therapy in Women With Uterine Fibroids or Endometriosis Who Are 18 to 50 Years of Age and at Risk for Pregnancy
Brief Title: Study of the Safety and Contraceptive Efficacy of Relugolix Combination Therapy in Women With Uterine Fibroids or Endometriosis Who Are at Risk for Pregnancy
Acronym: SERENE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma Switzerland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVT-601-050
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Contraception
Keywords: Relugolix; Estradiol; Norethindrone acetate; Uterine Fibroids; Endometriosis
MeSH Terms: conditions — Leiomyoma; Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Relugolix/E2/NETA (Experimental): Participants will receive relugolix combination therapy for 1 year (13 consecutive 28-day treatment cycles).
  Interventions: Drug: Relugolix Combination Therapy

INTERVENTIONS:
Drug: Relugolix Combination Therapy — Participants will receive orally 1 fixed-dose combination tablet (relugolix 40 mg/E2 1 mg/NETA 0.5 mg) once daily.
  Other Names: Myfembree

SUMMARY:
The purpose of this study is to assess the contraceptive efficacy of relugolix combination therapy.

DETAILED DESCRIPTION:
This is a single-arm, open-label, phase 3 study to assess the contraceptive efficacy of relugolix combination therapy (relugolix 40 milligrams [mg], estradiol [E2] 1 mg, and norethindrone acetate [NETA] 0.5 mg).

ELIGIBILITY:
Key Inclusion Criteria:

1. Is a premenopausal woman, 18 to 50 years of age.
2. Is at risk of pregnancy (that is, having heterosexual intercourse at least once per month) and is seeking contraception.
3. Has normal, regular menstrual cycles that are between 21 and 35 days in duration.
4. Has a diagnosis of uterine fibroids or endometriosis meeting either of the following criteria:

   1. Diagnosis of uterine fibroids by confirmation of ultrasound performed in the last 2 years and patient report of heavy menstrual bleeding affecting quality of life.
   2. Diagnosis of endometriosis and has had surgical or direct visualization (laparoscopy or laparotomy) and/or histopathologic confirmation of endometriosis, and the patient reports moderate, severe, or very severe pain during the most recent menses and/or during nonmenstrual portion of the cycle in the prior month
5. Is willing to use the study intervention as the sole method of contraception for 13 consecutive 28-day treatment cycles and does not intend to use any other form of contraception (for example, condoms).

Key Exclusion Criteria:

1. Is pregnant, or breastfeeding, or has breastfed in the last year.
2. Has a known history of infertility or sub-fertility.
3. Has presence or history of a venous thromboembolic event (for example, deep vein thrombosis, pulmonary embolism), an arterial thrombotic or thromboembolic event (for example, myocardial infarction, stroke, or peripheral arterial), or a transient ischemic attack, angina pectoris, or claudication.
4. Has a higher risk of arterial, venous thrombotic, or thromboembolic disorders.
5. Has a history of migraine with aura or focal neurological symptoms.
6. Has uncontrolled hypertension, diabetes with inadequate control, or multiple cardiovascular risk factors.
7. Has a history of clinically significant ventricular arrhythmias.
8. Has clinically significant liver disease, including active viral hepatitis or cirrhosis.
9. Has a history of pancreatitis associated with severe hypertriglyceridemia.
10. Has known human immunodeficiency virus (HIV) infection or high risk of contracting HIV.
11. Has a hepatic hemangioma or has a history of cholestasis with prior estrogen use or during pregnancy.
12. Has a serious contraindication to pregnancy (for example, a medical condition or use of chronic medication such as isotretinoin or thalidomide).
13. History of suicidal ideation or behavior, or confirmed "yes" to any question (with exception of non-suicidal self-injurious behavior, unless deemed as an unacceptable risk by the investigator) on the C-SSRS.
14. Has a bone mineral density Z-score ≤ -2.0 at lumbar spine, femoral neck, or total hip during the screening period.
15. Has a history of or currently has osteoporosis, or other metabolic bone disease, collagen vascular disease, chronic kidney disease (CKD) stage 3 or greater with glomerular filtration rate (GFR) < 60 mL/min/m2 using Modification of Diet in Renal Disease (MDRD) method, hyperparathyroidism, hyperprolactinemia, known pituitary adenoma, hyperthyroidism, anorexia nervosa, abnormal bone mineral metabolism (eg, hypophosphatemia), or low traumatic (fragility) fracture.
16. Has used chronic glucocorticoids that are oral, parenteral, inhaled (prednisone equivalents of ≥ 2.5 mg daily for ≥ 3 months) in 12 months prior to the study.
17. Has known BRCA mutation or other mutation associated with increased risk of breast cancer.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 1020 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Contraceptive Efficacy of Relugolix Combination Therapy as Assessed by the At-Risk Pearl Index (PI) | 13 consecutive 28-day treatment cycles
  The At-Risk PI is defined as the number of on treatment pregnancies per 100 women-years of treatment. The At-Risk PI will be calculated on the basis of cycles considered at-risk of pregnancy, that is, consecutive 28-day periods without use of any other contraceptive methods and with affirmed occurrence of vaginal intercourse. On-treatment pregnancies are pregnancies with an estimated conception date between the first day of study intervention intake up to and including 7 days after the last intake of study medication.

SECONDARY OUTCOMES:
Contraceptive Efficacy of Relugolix Combination Therapy as Assessed by the Modified At-Risk PI | 13 consecutive 28-day treatment cycles
  The Modified At-Risk PI is based on the number of on-treatment pregnancies occurring during cycles without any other contraceptive methods, regardless of occurrence of vaginal intercourse. On-treatment pregnancies are pregnancies with an estimated conception date between the first day of study intervention intake up to and including 7 days after the last intake of study medication.
Contraceptive Efficacy of Relugolix Combination Therapy as Assessed by the Gross PI | 13 consecutive 28-day treatment cycles
  The "typical use" contraceptive efficacy will be assessed using the Gross PI, based on the number of on-treatment pregnancies occurring during all cycles regardless of the use of other contraceptive methods, confirmed vaginal intercourse, or protocol compliance. On-treatment pregnancies are pregnancies with an estimated conception date between the first day of study intervention intake up to and including 7 days after the last intake of study medication.
Contraceptive Efficacy of Relugolix Combination Therapy as Assessed by the Method Failure PI | 13 consecutive 28-day treatment cycles
  The "perfect use" contraceptive efficacy will be assessed using the Method Failure PI, based on the number of on-treatment pregnancies occurring during cycles that are at risk and without major protocol deviations. On-treatment pregnancies are pregnancies with an estimated conception date between the first day of study intervention intake up to and including 7 days after the last intake of study medication.
Contraceptive Efficacy of Relugolix Combination Therapy as Assessed by the Cumulative 1-Year Pregnancy Rates | 13 consecutive 28-day treatment cycles
Incidence of Treatment-Emergent Adverse Events | 54 Weeks
Number of Participants Who Do Not Complete 13 Treatment Cycles | 13 consecutive 28-day treatment cycles
Percent Change in Bone Mineral Density from Baseline to 6 and 12 Months On-Treatment | 12 Months On-Treatment or EOT
  The percent change in bone mineral density will be measured from baseline to 6- and 12-months on treatment at the lumbar spine (L1-L4), total hip, and femoral neck.
Percent Change in Bone Mineral Density from Baseline an 12 Months On-Treatment (or EOT) to 6 and 12 Months Post-Treatment | 12 Months Post-Treatment Follow-Up
  The percent change in bone mineral density will be measured from baseline and 12-months on-treatment (or End-of-Treatment) to 6- and 12-months post-treatment at the lumbar spine (L1-L4), total hip, and femoral neck.

CONTACTS AND LOCATIONS:
Locations (94):
- United States (92):
  - Mobile, Mobile, Alabama
  - Chandler, Chandler, Arizona
  - Mesa, Mesa, Arizona
  - Peoria, Peoria, Arizona
  - Phoenix, Phoenix, Arizona
  - Burbank, Burbank, California
  - Canoga Park, Canoga Park, California
  - Encinitas, Encinitas, California
  - Gardena, Gardena, California
  - Lancaster, Lancaster, California
  - Long Beach, Long Beach, California
  - Palo Alto, Palo Alto, California
  - Sacramento, Sacramento, California
  - San Diego, San Diego, California
  - San Fernando, San Fernando, California
  - Valley Village, Valley Village, California
  - West Covina, West Covina, California
  - Aurora, Aurora, Colorado
  - Greenwood Village, Greenwood Village, Colorado
  - Washington, Washington D.C., District of Columbia
  - Aventura, Aventura, Florida
  - Boynton Beach, Boynton Beach, Florida
  - Davie, Davie, Florida
  - Deland, DeLand, Florida
  - Hialeah, Hialeah, Florida
  - Jacksonville, Jacksonville, Florida
  - Kissimmee, Kissimmee, Florida
  - Lake Worth, Lake Worth, Florida
  - Loxahatchee, Loxahatchee Groves, Florida
  - Margate, Margate, Florida
  - Miami, Miami, Florida
  - New Port Richey, New Port Richey, Florida
  - Orlando, Orlando, Florida
  - Panama City, Panama City, Florida
  - Sarasota, Sarasota, Florida
  - Atlanta, Atlanta, Georgia
  - College Park, College Park, Georgia
  - Columbus, Columbus, Georgia
  - Norcross, Norcross, Georgia
  - Sandy Springs, Sandy Springs, Georgia
  - Savannah, Savannah, Georgia
  - Smyrna, Smyrna, Georgia
  - Meridian, Meridian, Idaho
  - Nampa, Nampa, Idaho
  - Chicago, Chicago, Illinois
  - Brownsburg, Brownsburg, Indiana
  - Mishawaka, Mishawaka, Indiana
  - Shawnee, Shawnee, Kansas
  - Covington, Covington, Louisiana
  - Marrero, Marrero, Louisiana
  - Metairie, Metairie, Louisiana
  - New Orleans, New Orleans, Louisiana
  - Shreveport, Shreveport, Louisiana
  - Baltimore, Baltimore, Maryland
  - Towson, Towson, Maryland
  - Dearborn Heights, Dearborn Heights, Michigan
  - Detroit, Detroit, Michigan
  - Saginaw, Saginaw, Michigan
  - Jackson, Jackson, Mississippi
  - Saint Louis, St Louis, Missouri
  - Las Vegas, Las Vegas, Nevada
  - North Las Vegas, North Las Vegas, Nevada
  - Cherry Hill, Cherry Hill, New Jersey
  - Albuquerque, Albuquerque, New Mexico
  - New York, New York, New York
  - Durham, Durham, North Carolina
  - New Bern, New Bern, North Carolina
  - Raleigh, Raleigh, North Carolina
  - Winston-Salem, Winston-Salem, North Carolina
  - Minot, Minot, North Dakota
  - Columbus, Columbus, Ohio
  - Fairfield, Fairfield, Ohio
  - Franklin, Franklin, Ohio
  - Portland, Portland, Oregon
  - Philadelphia, Philadelphia, Pennsylvania
  - Myrtle Beach, Myrtle Beach, South Carolina
  - Summerville, Summerville, South Carolina
  - Chattanooga, Chattanooga, Tennessee
  - Memphis, Memphis, Tennessee
  - Austin, Austin, Texas
  - Beaumont, Beaumont, Texas
  - Dallas, Dallas, Texas
  - Fort Worth, Fort Worth, Texas
  - Houston, Houston, Texas
  - League City, League City, Texas
  - Pearland, Pearland, Texas
  - San Antonio, San Antonio, Texas
  - Salt Lake City, Salt Lake City, Utah
  - Annandale, Annandale, Virginia
  - Norfolk, Norfolk, Virginia
  - Bellevue, Bellevue, Washington
  - Seattle, Seattle, Washington
- Puerto Rico (2):
  - Cidra, Cidra
  - San Juan, San Juan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neblett MF 2nd, Stewart EA. Oral Gonadotropin-Releasing Hormone Antagonists for the Treatment of Uterine Leiomyomas. Obstet Gynecol. 2023 May 1;141(5):901-910. doi: 10.1097/AOG.0000000000005145. Epub 2023 Apr 5. PMID 37103532